CLINICAL TRIAL: NCT01153295
Title: "Functional Bowel Disorder. Investigation in General Practice"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Mejeribrugets ForskningsFond (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Luise Molenberg Begtrup, Doctor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MFF080408-1
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2008-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Irritable bowel syndrome; diagnosis; safety; Health related quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive diagnosis (Experimental): The diagnosis of IBS is based on the international ROME III criteria, few blod tests, and abscence of danger signals
  Interventions: Procedure: Clinical diagnosis based on symptom criteria
- Diagnosis of exclusion (Active Comparator): The diagnosis of IBS is based on normal extended blood tests, screening for celiac sprue and lactose intolerance, stool for ova and parasites and endoscopy with biopsy
  Interventions: Procedure: Diagnosis of exclusion

INTERVENTIONS:
Procedure: Clinical diagnosis based on symptom criteria — The diagnosis is based on ROME III criteria, abscence of danger signals and FBC, CRP
  Arms: Positive diagnosis
Procedure: Diagnosis of exclusion — The diagnosis is based on normal investigations involving endoscopy with biopsy, stool for ova and parasites, FBC, CRP, TSH, Ca, ALT, alanine aminotransferase; alkaline phosphatase, serum bilirubin, Screening for lactose and celiac sprue
  Arms: Diagnosis of exclusion

SUMMARY:
The study aims to investigate how to give the diagnosis of Irritable Bowel Syndrome.

The investigators compare two parallel groups of primary care patients, in the age of 18-50 years with gastrointestinal complaints where the GP suspects IBS. All included patients fulfil international diagnostic criteria (ROME III) and have no danger signals.

Group 1: The diagnosis is based on the diagnostic criteria and few blod tests Group 2: The diagnosis is a diagnosis of exclusion after investigations with extended blod tests, examination for milk- and gluten intolerance, stoll for ova and parasites and scopy of the intestine.

After receiving the diagnosis of Irritable bowel syndrome all patients are informed about the condition.

The investigators follow the patients for 1 year. The investigators hypothesis is that the two investigation programmes (group 1 and 2)are equal with respect to the patients´ quality of life, symptoms and satisfaction and also with respect to finding of organic diseases.

DETAILED DESCRIPTION:
Background: Two opposing approaches can be distinguished in establishing the diagnosis of Irritable Bowel Syndrome (IBS): IBS as a "diagnosis of exclusion" versus IBS as a syndromic condition on its own. In Denmark we have no consensus on how to establish the diagnosis, but must often GPs approach IBS as a diagnosis of exclusion. Guidelines from the United Kingdom and the United States recommend the second approach, where the diagnosis is given as a positive diagnosis based on symptom-based IBS criteria. We lack research on this area carried out under controlled circumstances and in primary care in Denmark.

Aim: To evaluate two investigation programmes for diagnosing IBS in primary care patients in Denmark. We want to compare the two programmes in relation to the effect on the patients´ symptoms, quality of life and satisfaction, and also the cost and safety when using the different programmes. Also we want to see how the GP´s understanding of IBS correlate with the IBS criteria (ROM I, II and III)

Methods: A randomised, non-blinded, controlled intervention study of two parallel groups.

The target group comprises people aged 18-50 years, who consult their GP with gastrointestinal complaints, where the GP suspects IBS and refers the patient to the study.

To be included in the study the patients have to fulfil the ROM III criteria and they may not have any alarm signals. Included patients are randomised to one of two different investigation programmes, where the diagnosis is given as:

1. A positive diagnosis, the diagnosis is based on the ROM III criteria and a few blood tests (FBC, CRP)
2. A diagnosis of exclusion, the diagnosis is given after normal investigation (extended blood tests, screening for celiac sprue and lactose intolerance, endoscopy)

The patients are followed by means of monthly letters, with questions about current GI symptoms, sick-leave days, visits at GPs, use of medication etc., and validated questionnaires at baseline, after 4 weeks, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill ROME III criteria
* age 18-50 years
* signed informed content

Exclusion Criteria:

* Danger signals (fever, anaemia, weightloss, blod in stools, predisposition for CRC or IBD)
* abnormal physical examination
* comorbidity
* abuse
* lacking ability to talk and understand danish
* pregnancy
* Performed endoscopy within the last 3 years
* For patients > 40 years. Changed bowel habits, with duration > 3 weeks, but < 1 year
* Age < 18 years and > 50 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | One year

SECONDARY OUTCOMES:
Findings of organic disease | one year
  We will look at the findings of organic disease (for example celiac disease or colorectal cancer) in the two investigation programes.

CONTACTS AND LOCATIONS:
Overall Officials: Ove B. Schaffalitzky de Muckadell, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Research Unit for General Practice, Department of gastroenterology, Odense University hospital, Odense, Odense, Denmark

REFERENCES:
- [Derived] Engsbro AL, Begtrup LM, Haastrup P, Storsveen MM, Bytzer P, Kjeldsen J, Schaffalitzky De Muckadell O, Jarbol DE. A positive diagnostic strategy is safe and saves endoscopies in patients with irritable bowel syndrome: A five-year follow-up of a randomized controlled trial. Neurogastroenterol Motil. 2021 Mar;33(3):e14004. doi: 10.1111/nmo.14004. Epub 2020 Oct 7. PMID 33029843
- [Derived] Begtrup LM, Engsbro AL, Kjeldsen J, Larsen PV, Schaffalitzky de Muckadell O, Bytzer P, Jarbol DE. A positive diagnostic strategy is noninferior to a strategy of exclusion for patients with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2013 Aug;11(8):956-62.e1. doi: 10.1016/j.cgh.2012.12.038. Epub 2013 Jan 26. PMID 23357491